CLINICAL TRIAL: NCT03217136
Title: A Phase 2, Randomized, Active Comparator-Controlled, Multicenter, Double-Blind Clinical Trial to Study the Safety and Efficacy of Ceftolozane/Tazobactam (MK-7625A) Plus Metronidazole Versus Meropenem in Pediatric Subjects With Complicated Intra-Abdominal Infection
Brief Title: MK-7625A Plus Metronidazole Versus Meropenem in Pediatric Participants With Complicated Intra-Abdominal Infection (cIAI) (MK-7625A-035)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7625A-035; MK-7625A-035 (Other: Merck); 2016-004820-41 (EudraCT Number)
Record Dates: First submitted 2017-07-12; First posted 2017-07-13 (Actual); Results first posted 2021-12-21 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Complicated Intra-Abdominal Infection
MeSH Terms: interventions — ceftolozane, tazobactam drug combination; Metronidazole; Meropenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ceftolozane/Tazobactam + Metronidazole (Experimental): Ceftolozane 20 mg/kg and tazobactam 10 mg/kg (maximum 1 g and 0.5 g/dose), plus metronidazole 10 mg/kg (maximum 1.5 g/day) administered intravenously (IV) every 8 to 12 hours for 5 to 14 days.
  Interventions: Drug: Ceftolozane/Tazobactam; Drug: Metronidazole
- Meropenem + Placebo for Metronidazole (Active Comparator): Meropenem 20 mg/kg (maximum 1 g/dose) plus placebo for Metronidazole administered IV every 8 hours for 5 to 14 days.
  Interventions: Drug: Meropenem; Drug: Placebo for Metronidazole

INTERVENTIONS:
Drug: Ceftolozane/Tazobactam — Ceftolozane 20 mg/kg (maximum 1 g) and tazobactam 10 mg/kg (maximum 0.5 g/dose) administered IV every 8 hours for between 5 to 14 days.
  Other Names: MK-7625A
  Arms: Ceftolozane/Tazobactam + Metronidazole
Drug: Metronidazole — Metronidazole 10 mg/kg (maximum 1.5 g/day) administered IV every 8 hours for between 5 to 14 days. Participants ≤ 28 days old, start with a loading dose of 15 mg/kg; then if ≤ 2 kg are dosed 7.5 mg/kg/ every 12 hours; or if > 2 kg are dosed 10 mg/kg every 8 hours.
  Arms: Ceftolozane/Tazobactam + Metronidazole
Drug: Meropenem — Meropenem 20 mg/kg (maximum 1 g/dose) administered IV every 8 hours for between 5 to 14 days.
  Other Names: MERREM
  Arms: Meropenem + Placebo for Metronidazole
Drug: Placebo for Metronidazole — Placebo for metronidazole administered IV every 8 hours for between 5 to 14 days.
  Arms: Meropenem + Placebo for Metronidazole

SUMMARY:
This study aims to evaluate the safety and tolerability of MK-7625A (ceftolozane/tazobactam) plus metronidazole, compared with that of meropenem in pediatric participants with cIAI.

ELIGIBILITY:
Inclusion Criteria:

* Has a legally acceptable representative who provides documented informed consent/assent for the trial.
* Aged from birth (defined as >32 weeks gestational age and ≥7 days postnatal) to <18 years of age.
* Require IV antibacterial therapy for the treatment of presumed or documented cIAI.
* Has an operative procedure for the current diagnosis and management of cIAI planned or completed within 24 hours of the first dose of an antibacterial drug. Note: Participants with a diagnosis of necrotizing enterocolitis are exempt and not required to have surgery planned or completed in order to be eligible.
* Has in compliance baseline intra-abdominal specimen collection.
* Is not of reproductive potential; but if of reproductive potential agrees to avoid becoming pregnant or impregnating a partner during screening, while receiving study treatment and for at least 30 days after the last dose of study treatment.
* Female of reproductive potential is not pregnant, and not planning to become pregnant within 30 days of the last day of treatment administration; and is nonlactating.

Exclusion Criteria:

* Is currently participating in or has participated in an interventional clinical trial with an investigational compound or device within 30 days prior to the first dose of study treatment in this current trial.
* Has previously participated in any trial of ceftolozane or ceftolozane/tazobactam or has enrolled previously in the current trial and been discontinued.
* Has a history of any moderate or severe hypersensitivity (e.g, anaphylaxis), allergic reaction, or other contraindication to any of the following: β-lactam antibiotics (e.g, penicillins, cephalosporins, and carbapenems), β-lactamase inhibitors (e.g, tazobactam, sulbactam, clavulanic acid, avibactam), or metronidazole.
* Has an IAI within the past 1 year prior to randomization known to be caused by a pathogen resistant to either IV study treatment.
* Has a concomitant infection at the time of randomization that requires non-study systemic antibacterial therapy in addition to IV study treatment or oral step-down therapy.
* Has received potentially therapeutic antibacterial therapy for a duration more than 24 hours during the 48 hours preceding the first dose of study treatment, unless is considered to be failing antibiotic therapy for cIAI.
* Has any of the following: a) intractable cIAI that the investigator anticipates would require more than 14 days of study treatment; b) abdominal wall abscess; c) small bowel obstruction; d) ischemic bowel disease without perforation; e) traumatic bowel perforation with surgery within 12 hours of perforation; f) perforation of gastroduodenal ulcers requiring surgery within 24 hours of perforation; g) suspected uncomplicated intra-abdominal infection (e.g, cholecystitis without rupture or extension beyond the gallbladder wall); h) acute suppurative cholangitis; i) infected necrotizing pancreatitis; j) pancreatic abscess.
* Has moderate or severe impairment of renal function.
* Has a seizure disorder or is anticipated to be treated with divalproex sodium or valproic acid during the course of study treatment.
* Is receiving, or is expected to receive, any prohibited medications.
* Has any rapidly progressing disease or immediately life-threatening illness, including acute hepatic failure, respiratory failure, or septic shock.
* Has an immunocompromising condition.
* Has a history of malignancy ≤5 years prior to signing informed consent.
* Is planning to receive suppressive/prophylactic antibiotics with gram-negative activity after completion of study treatment.

Ages: 7 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (50):
- United States (9):
  - Children's Hospital - Los Angeles ( Site 2508), Los Angeles, California
  - Children's Hospital of Orange County ( Site 2502), Orange, California
  - Rady Children's Hospital-San Diego ( Site 2505), San Diego, California
  - Baptist Medical Center/Wolfson Children's Hospital ( Site 2521), Jacksonville, Florida
  - Tufts Medical Center-Floating Hospital for Children ( Site 2516), Boston, Massachusetts
  - St. Louis Children's Hospital ( Site 2511), St Louis, Missouri
  - SUNY Upstate Medical University Hospital ( Site 2509), Syracuse, New York
  - Primary Children's Hospital ( Site 2500), Salt Lake City, Utah
  - Seattle Childrens Hospital ( Site 2510), Seattle, Washington
- Brazil (3):
  - Hospital Pequeno Principe ( Site 0200), Curitiba, Paraná
  - Inst de Medicina Integral Professor Fernando Figueira- IMIP ( Site 0201), Recife, Pernambuco
  - Hospital Tacchini ( Site 0203), Bento Gonçalves, Rio Grande do Sul
- Hungary (6):
  - PTE AOK Klinikai Kozpont ( Site 0805), Pécs, Baranya
  - SzSzBMK es Egyetemi Oktatokorhaz Josa Andras Oktatokorhaz ( Site 0804), Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Semmelweis Egyetem ( Site 0807), Budapest
  - Heim Pal Orszagos Gyermekgyogyaszati Intezet ( Site 0806), Budapest
  - Debreceni Egyetem Klinikai Kozpont ( Site 0801), Debrecen
  - SZTE Szent-Gyorgyi Albert Klinikai Kozpont ( Site 0802), Szeged
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kaunas ( Site 1001), Kaunas
  - Klaipedos Vaiku Ligonine ( Site 1000), Klaipėda
  - Vaiku Ligonine VU ligonines Santariskiu kliniku filialas ( Site 1002), Vilnius
- Malaysia (3):
  - Universiti Kebangsaan Malaya Medical Centre ( Site 1101), Cheras, Johor
  - Hospital Pulau Pinang ( Site 1102), George Town, Pulau Pinang
  - University Malaya Medical Centre. ( Site 1100), Kuala Lumpur
- Mexico (4):
  - Hospital del Nino y Adolescente Morelense ( Site 1204), Emiliano Zapata, Morelos
  - Instituto Tecnologico y de Estudios Superiores de Monterrey ( Site 1203), Monterrey, Nuevo León
  - Instituto Nacional de Pediatria ( Site 1201), Mexico City
  - Hospital Infantil de Mexico Federico Gomez ( Site 1202), Mexico City
- Romania (2):
  - Spit. Cl. de Urg. Copii Cluj Napoca ( Site 1703), Cluj-Napoca, Cluj
  - Spitalul Clinic de Urgenta pentru Copii "Louis Turcanu" Timi ( Site 1701), Timișoara, Timiș County
- Russia (4):
  - Chelyabinsk Regional Children Clinical Hospital ( Site 1802), Chelyabinsk, Chelyabinsk Oblast
  - Smolensk Regional Clinical Hospital ( Site 1800), Smolensk, Smolensk Oblast
  - Stavropol Regional Pediatric Clinical Hospital ( Site 1805), Stavropol, Stavropol Kray
  - Regional Childrens Clinical Hospital ( Site 1809), Vologda, Vologda Oblast
- South Africa (2):
  - Molotlegi Street ( Site 1901), Pretoria, Gauteng
  - Red Cross War Memorial Children's Hospital ( Site 1902), Cape Town, Western Cape
- Spain (4):
  - Hospital Clinico Universitario de Santiago ( Site 2001), Santiago de Compostela, A Coruña [La Coruña]
  - Institut Catala d Oncologia Hospital Germans Trias i Pujol ( Site 2004), Badalona, Barcelona
  - Hospital Universitario Sant Joan de Deu ( Site 2000), Esplugues de Llobregat, Barcelona
  - Hospital Universitario la Fe ( Site 2003), Valencia, Valenciana, Comunitat
- Turkey (Türkiye) (4):
  - Cukurova Uni Tip Fak Cocuk Saglıgı ve Hasta ABD ( Site 2200), Adana
  - Hacettepe Universitesi Tip Fakultesi Hastanesi ( Site 2201), Ankara
  - Eskisehir Osmangazi Unv. Tip Fakultesi ( Site 2202), Eskişehir
  - SBU Sariyer Hamidiye Etfal Egitim ve Arastirma Hastanesi ( Site 2203), Istanbul
- Ukraine (6):
  - SI Dnipropetrovsk Regional Children Clinical Hospital DOR ( Site 2452), Dnipro, Dnipropetrovsk Oblast
  - PI Kryvorizka city clinical hospital 8 ( Site 2458), Kryvyy Rig, Dnipropetrovsk Oblast
  - Ivano-Frankivsk Regional Children Clinical Hospital ( Site 2461), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - National Children Specialised Hospital OHMADYT MOH Ukraine ( Site 2459), Kyiv, Kyivska Oblast
  - Municipal Institution City Children s Clinical Hospital of Poltava City Council ( Site 2454), Poltava, Poltava Oblast
  - Vinnytsya Regional Children Clinical Hospital ( Site 2463), Vinnytsia, Vinnytsia Oblast

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Jackson CA, Newland J, Dementieva N, Lonchar J, Su FH, Huntington JA, Bensaci M, Popejoy MW, Johnson MG, De Anda C, Rhee EG, Bruno CJ. Safety and Efficacy of Ceftolozane/Tazobactam Plus Metronidazole Versus Meropenem From a Phase 2, Randomized Clinical Trial in Pediatric Participants With Complicated Intra-abdominal Infection. Pediatr Infect Dis J. 2023 Jul 1;42(7):557-563. doi: 10.1097/INF.0000000000003911. Epub 2023 Mar 29. PMID 37000942

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Paediatric participants were enrolled from 27 sites in 11 countries.
Groups:
- Meropenem: Meropenem 20 mg/kg (maximum 1 g/dose) plus placebo for metronidazole administered IV every 8 hours for 5 to 14 days.
Period: Overall Study
Arm/Group | Ceftolozane/Tazobactam + Metronidazole | Meropenem
Started | 71 | 23
Treated | 70 | 21
Completed | 67 | 20
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Site Randomized Participant in Error | 0 | 1
Not completed — Did Not Meet Criteria after Randomization | 0 | 1
Not completed — Dispensing Error | 1 | 0
Not completed — Withdrawal by Parent/Guardian | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceftolozane/Tazobactam + Metronidazole | Meropenem | Total
Number analyzed (Participants) | 71 | 23 | 94
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.7 (4.4) | 8.6 (3.6) | 8.7 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 15 | 38
  Male | 48 | 8 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 7 | 25
  Not Hispanic or Latino | 50 | 16 | 66
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 1 | 7
  White | 61 | 20 | 81
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing ≥1 Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered study treatment and which did not necessarily have to have a causal relationship with this treatment. The number of participants who experienced an AE is presented.
Time Frame: Up to approximately 75 days
Population: All randomized participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam + Metronidazole | Meropenem
Number analyzed (Participants) | 70 | 21
Participants | 56 | 13
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam + Metronidazole vs Meropenem; Difference in Percentage (C/T+MTZ minus MERO); Test type: Other — The Miettinen & Nurminen method was used; Difference in Percentage = 18.1, 95% CI 2-sided [-2.6 to 41.1]

2. Primary Outcome: Number of Participants Who Discontinued Study Therapy Due to AE(s)
Description: An AE was defined as any untoward medical occurrence in a participant administered study treatment and which did not necessarily have to have a causal relationship with this treatment. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximately 18 days
Population: All randomized participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane/Tazobactam + Metronidazole | Meropenem
Number analyzed (Participants) | 70 | 21
Participants | 2 | 0
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam + Metronidazole vs Meropenem; Difference in Percentage (C/T+MTZ minus MERO); Test type: Other — The Miettinen & Nurminen method was used; Difference in Percentage = 2.9, 95% CI 2-sided [-12.9 to 9.9]

3. Secondary Outcome: Percentage of Participants With a Clinical Response of "Cure" at the End of Treatment (EOT) Visit
Description: The percentage of participants who had a clinical outcome of "cure" at the time of the EOT visit is presented. The "cure" clinical outcome was defined as complete resolution or marked improvement in signs and symptoms of the complicated intra-abdominal infection (cIAI) or return to pre-infection signs and symptoms such that no further antibiotic therapy (intravenous or oral) or surgical or drainage procedure is required for treatment of the cIAI. Participants who were missing clinical response data were considered treatment failures.
Time Frame: Up to approximately 27 days
Population: All randomized participants who received any amount of study treatment. Participants were included in the IV study treatment group to which they were randomized, irrespective of what treatment they actually received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceftolozane/Tazobactam + Metronidazole | Meropenem
Number analyzed (Participants) | 70 | 21
Percentage of participants | 80.0 [69.18 to 87.70] | 95.2 [77.33 to 99.15]
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam + Metronidazole vs Meropenem; Difference in Percentage (C/T+MTZ minus MERO); Test type: Other — The difference in percentage was based on the Miettinen & Nurminen method stratified by age group with Cochran-Mantel-Haenszel (CMH) weights. If there was a zero count in any class of the stratum, the groups with the lower count were pooled with its near age group stratum in the model; Difference in Percentage = -14.3, 95% CI 2-sided [-26.67 to 4.93]

4. Secondary Outcome: Percentage of Participants With a Clinical Response of "Cure" at the Test of Cure (TOC) Visit
Description: The percentage of participants who had a clinical outcome of "cure" at the time of the TOC visit is presented. The "cure" clinical outcome was defined as complete resolution or marked improvement in signs and symptoms of the complicated intra-abdominal infection (cIAI) or return to pre-infection signs and symptoms such that no further antibiotic therapy (intravenous or oral) or surgical or drainage procedure is required for treatment of the cIAI. Participants who were missing clinical response data were considered treatment failures.
Time Frame: Up to approximately 39 days
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceftolozane/Tazobactam + Metronidazole | Meropenem
Number analyzed (Participants) | 70 | 21
Percentage of participants | 80.0 [69.18 to 87.70] | 100.0 [84.54 to 100.0]
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam + Metronidazole vs Meropenem; Difference in Percentage (C/T+MTZ minus MERO); Test type: Other — [test comment as in outcome 3, analysis 1]; Difference in Percentage = -19.1, 95% CI 2-sided [-30.18 to -2.89]

5. Secondary Outcome: Percentage of Participants With Microbiological Eradication at the EOT Visit
Description: The percentage of participants who achieved either eradication or presumed eradication of each baseline infecting pathogen by the time of the EOT visit is presented. Eradication was defined as absence of the baseline pathogen(s) in a postbaseline specimen appropriately obtained from the original site of infection. Presumed eradication was defined as absence of material to culture in a participant who is assessed as having partial improvement, or clinical cure. In the event of multiple baseline pathogens, the least favorable microbiological response from all possible baseline pathogens was used.
Time Frame: Up to approximately 27 days
Population: All randomized participants who received any amount of study treatment and had at least 1 pathogen identified from the baseline intra-abdominal culture, regardless of susceptibility to study treatment. Participants were included in the IV study treatment group to which they were randomized, irrespective of what treatment they actually received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceftolozane/Tazobactam + Metronidazole | Meropenem
Number analyzed (Participants) | 63 | 19
Percentage of participants | 84.1 [73.19 to 91.14] | 94.7 [75.36 to 99.06]
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam + Metronidazole vs Meropenem; Difference in Percentage (C/T+MTZ minus MERO); Test type: Other — [test comment as in outcome 3, analysis 1]; Difference in Percentage = -11.2, 95% CI 2-sided [-23.66 to 9.61]

6. Secondary Outcome: Percentage of Participants With Microbiological Eradication at the TOC Visit
Description: The percentage of participants who achieved either eradication or presumed eradication of each baseline infecting pathogen by the time of the TOC visit is presented. Eradication was defined as absence of the baseline pathogen(s) in a postbaseline specimen appropriately obtained from the original site of infection. Presumed eradication was defined as absence of material to culture in a participant who is assessed as having partial improvement, or clinical cure. In the event of multiple baseline pathogens, the least favorable microbiological response from all possible baseline pathogens was used.
Time Frame: Up to approximately 39 days
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceftolozane/Tazobactam + Metronidazole | Meropenem
Number analyzed (Participants) | 63 | 19
Percentage of participants | 84.1 [73.19 to 91.14] | 100 [83.18 to 100.00]
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam + Metronidazole vs Meropenem; Difference in Percentage (C/T+MTZ minus MERO); Test type: Other — [test comment as in outcome 3, analysis 1]; Difference in Percentage = -16.3, 95% CI 2-sided [-27.59 to 1.39]

ADVERSE EVENTS:
Time Frame: Up to approximately 75 days
Description: Deaths are counted in the population of all randomized participants. Serious adverse events and non-serious adverse events are reported for all randomized participants who received any amount of study treatment.
Arm/Group | Ceftolozane/Tazobactam + Metronidazole | Meropenem
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/23
Serious Adverse Events (participants affected / at risk) | 8/70 | 0/21
Other Adverse Events (participants affected / at risk) | 46/70 | 10/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftolozane/Tazobactam + Metronidazole (N=70) | Meropenem (N=21)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftolozane/Tazobactam + Metronidazole (N=70) | Meropenem (N=21)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 6 (6) | 1 (1)
Tachycardia (Cardiac disorders) | 5 (5) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (8) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 13 (14) | 5 (5)
Vomiting (Gastrointestinal disorders) | 7 (8) | 1 (1)
Pyrexia (General disorders) | 9 (10) | 3 (7)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (4)
Incision site pain (Injury, poisoning and procedural complications) | 7 (7) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 1 (1)
Platelet count increased (Investigations) | 5 (5) | 2 (2)
Hypertension (Vascular disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/36/NCT03217136/Prot_SAP_000.pdf